CLINICAL TRIAL: NCT01689831
Title: Dose Comparison Study of Tuberculin Purified Protein Derivative (PPD)With Standard Tuberculin Purified Protein Derivative.
Brief Title: Dose Study of Tuberculin Purified Protein Derivative (JHP/Dose)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: JHP Pharmaceuticals LLC (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: JHP - 42023
Record Dates: First submitted 2012-07-03; First posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Tuberculosis Infection
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aplisol, potency determination (Experimental): To confirm the potency of Aplisol formulated with newly produced Tuberculin PPD compared to PPD-S2 standard.
  Interventions: Biological: To confirm the potency of Aplisol formulated with newly produced Tuberculin PPD compared to PPD-S2 standard.; Biological: Reactivity of Aplisol compared to reference standard PPD-S2.
- Reference standard PPD-S2, reference (Active Comparator): Reactivity of Aplisol compared to reference standard PPD-S2.
  Interventions: Biological: To confirm the potency of Aplisol formulated with newly produced Tuberculin PPD compared to PPD-S2 standard.; Biological: Reactivity of Aplisol compared to reference standard PPD-S2.

INTERVENTIONS:
Biological: To confirm the potency of Aplisol formulated with newly produced Tuberculin PPD compared to PPD-S2 standard. — Comparison of different dosages of Aplisol PPD relative to reference standard PPD-S2.
Biological: Reactivity of Aplisol compared to reference standard PPD-S2. — Reference standard PPD-S2 formulated to contain different dose concentrations.
  Other Names: Reference standard PPD-S2.

SUMMARY:
Dose comparison study of tuberculin purified protein derivative (PPD)Aplisol with the standard tuberculin purified derivative (PPD-S2).

DETAILED DESCRIPTION:
JHP proposes to demonstrate clinical comparability of Aplisol formulated from the new Tuberculin PPD drug substance to the standard PPD-S2.

ELIGIBILITY:
Inclusion Criteria:

1. Males or nonpregnant females age 18 to 60 years
2. Documented PPD reactivity of 5 to 21 mm in the past, documented in a medical record. Self-reported PPD reactivity will be accepted if medical records cannot be obtained.
3. Give written informed consent to participate
4. Generally healthy, as determined by medical history and targeted physical examination, if indicated
5. Possess 2 forearms that are free of burns, scars, eczema, or any physical deformity, which could impair injection of study preparation or the readings of the injections
6. Comprehension of the study requirements; expressed availability for the required study period, including readings at the nominal time points of 48 and 72 hours

Exclusion Criteria:

1. Prior PPD test within the past 30 days
2. Subject is of childbearing potential and unable to use contraceptives; is planning pregnancy; is pregnant or lactating
3. History of anaphylactic reaction, severe positive tuberculin reaction (eg, ulceration, necrosis) or other severe reaction to PPD in the past
4. Subject received a Bacillus Calmette-Guérin (BCG) vaccination in the past, or was born or lived outside the US as a child and is uncertain of his/her BCG vaccination status
5. Presence of conditions that may suppress TST reactivity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Confirm the potency of Aplisol equipotent to PPD-S2. | 72 hours

SECONDARY OUTCOMES:
Assess tolerability of Aplisol with new tuberculin PPD | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center at Tyler, Tyler, Texas, United States